CLINICAL TRIAL: NCT00652522
Title: Atrial Fibrillation Management in Congestive Heart Failure With Ablation
Acronym: AMICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AF06003AF
Record Dates: First submitted 2008-03-20; First posted 2008-04-03 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Persistent Atrial Fibrillation; Heart Failure; ICD
Keywords: AF ablation; Pulmonary vein isolation(PVI); reduced LV ejection fraction; symptomatic atrial fibrillation; persistent AF
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Best Medical Treatment, ICD/CRT implant
  Interventions: Device: ICD/CRT implant; Other: Best Medical Treatment
- B (Experimental): AF Ablation, ICD/CRT implant
  Interventions: Device: ICD/CRT implant; Procedure: AF ablation

INTERVENTIONS:
Device: ICD/CRT implant — Implantation of a ICD/ CRT device if not yet implanted
  Other Names: ICDs/ CRT-Ds: All St. Jude Medical device; RA, RV and LV leads: St. Jude Medical CE-marked leads recommended
Procedure: AF ablation — Atrial Fibrillation ablation by pulmonary vein isolation
  Other Names: Catheters: St. Jude Medical CE-marked catheters recommended; NavX system for 3D mapping
  Arms: B
Other: Best Medical Treatment — Best medical treatment according to current guidelines for Management of Patients with Atrial Fibrillation and for Management of Chronic Heart Failure.
  Other Names: Conventional rate or rhythm control according valid guidelines
  Arms: A

SUMMARY:
It is the purpose of the study to show the benefit of the endocardial catheter ablation by pulmonary vein isolation in patients with persistent or longstanding persistent atrial fibrillation, low LVEF and requiring ICD or CRT-D therapy compared to the best medical treatment with antiarrhythmic drugs.

DETAILED DESCRIPTION:
Atrial fibrillation is the most common sustained cardiac arrhythmia affecting 5% of people older than 65 years. It is associated with a 5 times increase of the risk of stroke in patients who are not receiving anticoagulant therapy and a doubling of the rate of death in all patients.

Congestive heart failure (CHF) and atrial fibrillation (AF) often co-exist, where one condition is promoting the development of the other and worsens its condition.

It is the purpose of the study to show the benefit of the endocardial catheter ablation by pulmonary vein isolation in patients with persistent (for a minimum of 1 week to a maximum of 1 year duration) or longstanding persistent (for a minimum of 1 year to a maximum of 4 years) atrial fibrillation, low LVEF (<=35%) and requiring ICD or CRT-D therapy compared to the best medical treatment with antiarrhythmic drugs.

Patients meeting the inclusion and exclusion criteria will be randomized in a 1:1 fashion in an unblinded, parallel arm treatment format to either drug therapy (directed at rate or rhythm control) or catheter ablation.

All therapies will be established and optimized in a 3 month treatment initiation phase (Blanking Period) starting with randomization. For all morbidity and mortality end-points, intention-to-treat analysis will begin at randomization. Efficacy with respect to AF treatment will be established for long-term follow up beginning after 3-month initiation phase.

Improvement of LVEF within 12 month is the primary endpoint of this study. The transthoracic echocardiographic (TTE) assessment at enrollment, discharge and 12 months follow-up follows a standardized protocol. The assessments are analyzed, calculated and expressed by an independent Core Lab.

ELIGIBILITY:
Inclusion Criteria:

* Having signed and dated Patient Informed Consent
* Having an indication for ICD or CRT-D therapy as indicated by current valid guidelines or having been implanted with an ICD or CRT-D
* Symptomatic atrial fibrillation (persistent AF (for a minimum of 1 week to a maximum of 1 year) or longstanding persistent AF (for a minimum of 1 year to a maximum of 4 years)) irrespective of the duration of paroxysmal AF
* Ejection fraction ≤ 35% as assessed by transthoracic echocardiography
* Left atrial diameter of less than 60 mm in parasternal diameter during transthoracic echocardiographic study
* ECG documentation of atrial fibrillation (ECG, Holter, event recorders, etc) related to symptomatic episodes
* Having typical symptoms of heart failure NYHA II - III
* Patients > 30 days under optimal medical treatment for heart failure and CRT therapy in case of a pre-implanted CRT-D device
* Age 18 - 75 years
* Willing to participate in randomized trial
* Willing and able to participate in 12 months follow-up period

Exclusion Criteria:

* Longstanding persistent (> 4 years history) or paroxysmal atrial fibrillation
* Having a previously implanted pacemaker
* Having underlying valvular heart disease unless the disease has been corrected
* Patients with acute myocardial infarction
* Patients who have had previous pulmonary vein isolation procedures
* Patients with atrial fibrillation secondary to a reversible cause
* Known presence of intracardiac or other thrombi
* Pregnant females or those of child bearing potential who have not had a negative pregnancy test within 48 hours before treatment
* Patients with other medical condition (i.e., cancer, alcoholism, drug abuse) that may cause the patient to be non-compliant with the protocol, confound the data interpretation or is associated with limited life-expectancy (i.e., less than one year)
* History of bleeding diathesis or suspected pro-coagulant state
* Contraindication to anticoagulation therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (LVEF) by transthoracic echocardiography (TTE) | 12months
  evaluated by Core Lab

SECONDARY OUTCOMES:
Recurrence of atrial tachyarrhythmia | 9 months
  diagnosed by daily ECG via ECG-recording card
Exercise capacity in 6 min walk test | 12 months
Quality of life | 12 months
  assessed by Minnesota Quality of Life Questionnaire
AF burden | 9 months
  assessed by ICD/CRT-D device memory in SJM devices
Adverse events | 12 months
Mortality | 12 months
Number of adequate and inadequate ICD interventions | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Heinz Kuck, Prof., Principal Investigator — Asklepios Klinik St. Georg - Hamburg
Locations (16):
- Germany (14):
  - Herz- und Gefaesszentrum Bad Bevensen, Bad Bevensen
  - Universitäts-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen
  - Kerckhoff-Klinik gGmbH, Bad Nauheim
  - Universitätsmedizin Berlin - Charité Campus Virchow-Klinikum (CVK), Berlin
  - Herzzentrum Dresden, Dresden
  - Asklepios Klinik St. Georg, Hamburg
  - Universitäres Herzzentrum Hamburg GmbH / UKE, Hamburg
  - Klinikum der Ruprecht-Karls-Universität Heidelberg, Heidelberg
  - Klinikum Ingolstadt GmbH, Ingolstadt
  - Herzzentrum Leipzig GmbH, Leipzig
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - Klinikum Großhadern der Ludwig-Maximilians-Universität, München
  - Herzzentrum am Universitätsklinikum Münster, Münster
  - St. Adolf-Stift Reinbek, Reinbek
- Semmelweis University, Budapest, Hungary
- Hospital Universitari Clinic, Barcelona, Spain

REFERENCES:
- [Derived] Kuck KH, Merkely B, Zahn R, Arentz T, Seidl K, Schluter M, Tilz RR, Piorkowski C, Geller L, Kleemann T, Hindricks G. Catheter Ablation Versus Best Medical Therapy in Patients With Persistent Atrial Fibrillation and Congestive Heart Failure: The Randomized AMICA Trial. Circ Arrhythm Electrophysiol. 2019 Dec;12(12):e007731. doi: 10.1161/CIRCEP.119.007731. Epub 2019 Nov 25. PMID 31760819